CLINICAL TRIAL: NCT00235716
Title: CSP #546 - A Randomized, Clinical Trial of Vitamin E and Memantine in Alzheimer's Disease (TEAM-AD)
Brief Title: A Randomized, Clinical Trial of Vitamin E and Memantine in Alzheimer's Disease
Acronym: TEAM-AD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Forest Laboratories (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 546
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; clinical trial; randomized controlled trial; alpha-tocopherol; vitamin E; Namenda; memantine
MeSH Terms: conditions — Alzheimer Disease | interventions — alpha-Tocopherol; Vitamin E; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): 2,000 IU per day of dl-alpha-tocopherol plus placebo for memantine
  Interventions: Drug: dl-alpha-tocopherol
- Arm 2 (Experimental): 20 mg per day of memantine plus placebo for dl-alpha-tocopherol
  Interventions: Drug: Memantine
- Arm 3 (Experimental): Combination of 2,000 IU per day of dl-alpha-tocopherol and 20 mg per day of memantine
  Interventions: Drug: dl-alpha-tocopherol; Drug: Memantine
- Arm 4 (Placebo Comparator): Matching placebos for dl-alpha-tocopherol and memantine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dl-alpha-tocopherol — Alpha-tocopherol will be given as an oral dose of 1000 IU twice a day (morning and evening). The form of vitamin E that will be used in this study will be hard gel capsules of dl-alpha-tocopheryl acetate ("synthetic") vitamin E.
  Other Names: Vitamin E
  Arms: Arm 1
Drug: Memantine — A moderate-affinity NMDA antagonist. Memantine will be titrated over four weeks to a maintenance dose of 10 mg twice a day. During week 1 patients will take one 5-mg memantine tablet in the morning. During week 2 patients will take one 5-mg memantine tablet in the morning and one in the evening. During week 3 patients will take two 5-mg memantine tablets in the morning and one 5-mg tablet in the evening. Beginning with week 4, participants will take four 5-mg tablets daily, two in the morning and two in the evening.
  Other Names: Namenda (R)
  Arms: Arm 2
Drug: dl-alpha-tocopherol — Alpha-tocopherol will be given as an oral dose of 1000 IU twice a day (morning and evening). The form of vitamin E that will be used in this study will be hard gel capsules of dl-alpha-tocopheryl acetate ("synthetic") vitamin E.
  Other Names: Vitamin E
  Arms: Arm 3
Drug: Memantine — A moderate-affinity NMDA antagonist. Memantine will be titrated over four weeks to a maintenance dose of 10 mg twice a day. During week 1 patients will take one 5-mg memantine tablet in the morning. During week 2 patients will take one 5-mg memantine tablet in the morning and one in the evening. During week 3 patients will take two 5-mg memantine tablets in the morning and one 5-mg tablet in the evening. Beginning with week 4, participants will take four 5-mg tablets daily, two in the morning and two in the evening.
  Other Names: Namenda (R)
  Arms: Arm 3
Drug: Placebo — Matching placebos for dl-alpha-tocopherol and memantine.
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine whether alpha-tocopherol, memantine (Namenda), or the combination will significantly delay clinical progression in mild to moderately demented patients with Alzheimer's disease compared to placebo.

DETAILED DESCRIPTION:
Abstract: Alzheimer's disease (AD), a neurodegenerative disorder resulting in cognitive loss, behavioral problems, and functional decline, is characterized by well-established and well-known neuropathological changes in the brain. Cognitive deficits and behavioral symptoms are thought to be due to cholinergic neuronal degeneration and loss associated with oxidative stress and inflammatory responses.

Current therapeutic strategies include efforts to

1. enhance cholinergic neuronal function,
2. promote neuroprotective effects, and
3. block pathologic activity of excessive glutamate with a moderate-affinity NMDA antagonist.

A combination of pharmacological therapies directed at simultaneously improving neuronal function and neuroprotection would presumably be more effective than either treatment alone.

To test this hypothesis, this study will examine the efficacy of drug treatment with a combination of

1. any of three FDA approved cholinesterase inhibitors that facilitates central acetylcholine neurotransmission (donepezil, rivastigmine, galantamine);
2. alpha-tocopherol, a fat soluble vitamin that has been shown to slow the rate of progression of AD, presumably through neuroprotective mechanism that reduces oxidative stress; and
3. memantine, a moderate-affinity NMDA antagonist that blocks excessive stimulation of NMDA receptors by glutamate. CSP#546 will be a double-blind, placebo-controlled, randomized, clinical trial to assess the efficacy of adding alpha-tocopherol, memantine, and the combination for the treatment of functional decline in mild-to-moderately demented patients with Alzheimer's disease (MMSE 12-26) who are currently taking an acetylcholinesterase inhibitor (AchEI).

Eligible Veterans will be randomly assigned to either

1. 2,000 IU/d of alpha-tocopherol plus memantine placebo,
2. 20 mg/d of memantine (Namenda) plus alpha-tocopherol placebo,
3. 2,000 IU/d of alpha-tocopherol plus 20 mg/d of memantine, or
4. alpha-tocopherol placebo plus memantine placebo.

The primary outcome for the study will be progression of AD as measured by the Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS/ADL) inventory. The ADCS/ADL inventory is an established outcome measure that was designed to assess functional capacity over a broad range of dementia severity and to be sensitive in measuring dementia progression. Secondary outcome measures will include the following five instruments: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) (cognition), MMSE (cognition), The Dependence Scale (function), Neuropsychiatric Inventory (NPI) (behavior), and Caregiver Activity Survey (CAS) (caregiver time). Outcomes and safety assessments will be obtained at baseline and every six months. The target sample size for the trial will be 620 patients (210 per treatment arm). This sample size will provide 90% power to detect a 4-point mean treatment difference in the ADCS/ADL inventory by the end of the average follow-up period, adjusted for losses. The effects to be detected are modest and translate into a 17.7% reduction in the annual rate of decline with each therapy given alone, and if the effects are additive, an approximate 35% reduction for combined therapy. These effects are equivalent to slowing the rate of progression of the disease by nearly 6 months for monotherapy and 12 months for combined therapy. To achieve the target sample size, Veterans will be recruited over a 3-year period with an estimated minimum follow-up of 1 year and a maximum of 4 years. A total of 10 to 15 VA sites will be established to enroll an average of one Veteran every 2 weeks. CSP#546 is designed to assess both a clinically and economically important treatment effect. If the study definitely determined that alpha-tocopherol, memantine, or the combination delays the progression of AD, the study would be tremendously valuable in reducing the financial and emotional costs of the disease in the VA and U.S. as a whole.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of possible or probable Alzheimer's disease (NINCDS-ADRDA)
2. Presence of a caregiver (friend or relative) who can assume responsibility for medication compliance, can accompany the patient to all visits, and rate patient's condition
3. Written informed consent from both the patient (or surrogate) and caregiver
4. An MMSE score between 12 and 26 inclusive
5. Administration of a maintenance dosage of donepezil (5-10mg/d), rivastigmine (6-12mg/d) or rivastigmine (Exelon) patch (4.6 mg or 9.5 mg), galantamine or galantamine ER (16-24mg/d) for a minimum of 4 weeks prior to randomization
6. Agreement not to take vitamin E supplements and/or memantine outside of the study (daily multivitamin is permitted containing up to 100 IU alpha-tocopherol)

Exclusion Criteria:

1. A non-Alzheimer primary dementia (e.g., vascular dementia, Lewy body dementia, fronto-temporal dementia, vitamin B-12 deficiency, hypothyroidism)
2. Current major depression, delirium, alcohol or psychoactive substance abuse or dependency, schizophrenia, or delusional disorder as defined by DSM-IV
3. Presence of any uncontrolled systemic illness that would interfere with participation in the study or a life expectancy of less than one year
4. Pregnant or intention to become pregnant
5. Enrollment in another interventional clinical trial
6. Current prescription with more than one AChE inhibitor
7. Current prescription for warfarin
8. Use of vitamin E supplements in the past 2 weeks
9. Use of memantine in the past 4 weeks or known intolerance
10. Estimated creatinine clearance less than 5ml/min (Cockcroft-Gault formula)
11. Use of amantadine in the past 2 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2007-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Dysken, Study Chair — Minneapolis Veterans Affairs Medical Center
Locations (14):
- United States (13):
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - VA Medical Center, Miami, Miami, Florida
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - Salisbury VAMC, Salisbury, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Background] Dysken MW, Guarino PD, Vertrees JE, Asthana S, Sano M, Llorente M, Pallaki M, Love S, Schellenberg GD, McCarten JR, Malphurs J, Prieto S, Chen P, Loreck DJ, Carney S, Trapp G, Bakshi RS, Mintzer JE, Heidebrink JL, Vidal-Cardona A, Arroyo LM, Cruz AR, Kowall NW, Chopra MP, Craft S, Thielke S, Turvey CL, Woodman C, Monnell KA, Gordon K, Tomaska J, Vatassery G. Vitamin E and memantine in Alzheimer's disease: clinical trial methods and baseline data. Alzheimers Dement. 2014 Jan;10(1):36-44. doi: 10.1016/j.jalz.2013.01.014. Epub 2013 Apr 11. PMID 23583234
- [Result] Dysken MW, Sano M, Asthana S, Vertrees JE, Pallaki M, Llorente M, Love S, Schellenberg GD, McCarten JR, Malphurs J, Prieto S, Chen P, Loreck DJ, Trapp G, Bakshi RS, Mintzer JE, Heidebrink JL, Vidal-Cardona A, Arroyo LM, Cruz AR, Zachariah S, Kowall NW, Chopra MP, Craft S, Thielke S, Turvey CL, Woodman C, Monnell KA, Gordon K, Tomaska J, Segal Y, Peduzzi PN, Guarino PD. Effect of vitamin E and memantine on functional decline in Alzheimer disease: the TEAM-AD VA cooperative randomized trial. JAMA. 2014 Jan 1;311(1):33-44. doi: 10.1001/jama.2013.282834. PMID 24381967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated in August, 2007 and concluded in March, 2012. Enrollment took place at 14 VA medical centers.
Groups:
- Vitamin E: Alpha-tocopherol (vitamin E in the form of dl-alpha-tocopheryl acetate), 2000 international units (IU) per day, taken as one 1000 IU hard-gelatin, liquid-filled capsules twice a day plus matching memantine placebos.
- Memantine (Namenda): Memantine 20 mg per day, titrated over four weeks to a maintenance dosage of 10 mg pills taken twice a day plus matching vitamin E placebo.
- Vitamin E + Memantine: 2000 IU of Alpha-tocopherol (vitamin E) per day plus 20 mg memantine per day.
- Placebo: Matching placebo pills for vitamin E and memantine
Period: Overall Study
Arm/Group | Vitamin E | Memantine (Namenda) | Vitamin E + Memantine | Placebo
Started | 152 | 155 | 154 | 152
Completed | 90 | 88 | 89 | 90
Not Completed | 62 | 67 | 65 | 62
Not completed — Death | 26 | 39 | 32 | 31
Not completed — Withdrawal by Subject | 23 | 19 | 17 | 18
Not completed — Lost to Follow-up | 12 | 7 | 14 | 10
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E | Memantine (Namenda) | Vitamin E + Memantine | Placebo | Total
Number analyzed (Participants) | 152 | 155 | 154 | 152 | 613
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.6 (7.2) | 78.8 (7.2) | 78.3 (7.0) | 79.4 (7.0) | 78.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 3 | 19
  Male | 146 | 149 | 150 | 149 | 594
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 15 | 19 | 66
  Not Hispanic or Latino | 135 | 140 | 139 | 133 | 547
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 21 | 21 | 18 | 20 | 80
  White | 130 | 132 | 136 | 131 | 529
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 152 | 155 | 154 | 152 | 613
Education [Number; unit: participants]
  <High School Graduation | 41 | 41 | 26 | 29 | 137
  High School Graduation | 46 | 48 | 57 | 56 | 207
  Some College | 27 | 38 | 37 | 33 | 135
  College Graduation or Advanced Degree | 38 | 28 | 34 | 34 | 134
Apolipoprotein E ε4 status [Number; unit: participants] — Data collected through genetic sub-study with separate informed consent.
  participants
    Non-carriers | 47 | 48 | 59 | 55 | 209
    One ε4 allele | 39 | 44 | 44 | 38 | 165
    Two ε4 alleles | 10 | 13 | 8 | 10 | 41
    Not Tested | 56 | 50 | 43 | 49 | 198
Concomitant Medications Acetylcholinesterase Inhibitors (AChEI) [Number; unit: participants]
  Donepezil | 104 | 100 | 100 | 96 | 400
  Galantamine | 43 | 47 | 49 | 55 | 194
  Rivastigmine | 5 | 8 | 4 | 1 | 18
  None | 0 | 0 | 1 | 0 | 1
Weeks from AChEI Initiation to Randomization [Number; unit: participants]
  ≤ 12 weeks | 46 | 36 | 49 | 37 | 168
  > 12 weeks | 105 | 119 | 104 | 115 | 443
  Missing | 1 | 0 | 1 | 0 | 2
Alzheimer's Disease Cooperative Study/Activities of Daily Living Inventory [Mean (Standard Deviation); unit: units on a scale] | 56.6 (14.9) | 57.3 (14.2) | 56.4 (14.0) | 56.8 (13.7) | 56.8 (14.2)
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] | 21.3 (3.3) | 20.8 (3.8) | 21.3 (3.4) | 20.8 (3.8) | 21.0 (3.6)
Alzheimer's Disease Assessment Scale - Cognitive portion [Mean (Standard Deviation); unit: units on a scale] | 18.5 (8.8) | 19.5 (7.9) | 18.0 (8.4) | 19.1 (8.4) | 18.8 (8.4)
Neuropsychiatric Inventory [Mean (Standard Deviation); unit: units on a scale] | 12.2 (13.3) | 12.1 (13.1) | 12.3 (13.3) | 13.5 (14.2) | 12.5 (13.4)
Caregiver Activity Survey [Mean (Standard Deviation); unit: hours per day] | 7.3 (14.3) | 6.7 (9.0) | 6.6 (10.5) | 6.5 (9.2) | 6.8 (10.9)
Dependence Scale [Number; unit: participants] — Higher the level the more dependence / less independence.
  participants
    Level 0 | 5 | 6 | 8 | 3 | 22
    Level 1 | 8 | 6 | 8 | 5 | 27
    Level 2 | 85 | 91 | 80 | 79 | 335
    Level 3 | 31 | 35 | 31 | 37 | 134
    Level 4 | 4 | 7 | 10 | 8 | 29
    Level 5 | 19 | 10 | 17 | 20 | 66

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS/ADL) Inventory Change From Baseline
Description: The primary outcome of the study was the Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS/ADL) Inventory. The ADCS/ADL Inventory is designed to assess functional abilities to perform activities of daily living in Alzheimer patients with a broad range of dementia severity. The total score ranges from 0 to 78 with higher scores indicating greater abilities. Outcome analysis is average least square means change from baseline.
Time Frame: 6, 12, 18, 24, 30, 36, 42 and 48 months minus baseline
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Memantine: Memantine 20 mg per day, titrated over four weeks to a maintenance dosage of 10 mg pills taken twice a day plus matching vitamin E placebo.
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 140 | 142 | 139 | 140
units on a scale
  6 months minus baseline | -1.72 (0.95) | -2.40 (0.94) | -2.78 (0.96) | -4.52 (0.95)
  12 months minus baseline | -4.29 (1.20) | -6.99 (1.21) | -6.60 (1.21) | -8.11 (1.23)
  18 months minus baseline | -8.01 (1.40) | -9.32 (1.42) | -7.98 (1.41) | -10.21 (1.43)
  24 months minus baseline | -11.88 (1.66) | -14.06 (1.70) | -12.82 (1.68) | -16.18 (1.74)
  30 months minus baseline | -15.84 (1.94) | -18.30 (1.97) | -15.66 (1.97) | -19.67 (2.06)
  36 months minus baseline | -19.71 (2.34) | -18.78 (2.43) | -18.89 (2.32) | -24.82 (2.51)
  42 months minus baseline | -25.30 (2.57) | -23.48 (2.65) | -23.44 (2.52) | -28.13 (2.76)
  48 months minus baseline | -26.55 (3.11) | -24.60 (3.18) | -29.25 (3.08) | -27.55 (3.38)
  Average change from baseline | -13.81 (1.11) | -14.98 (1.10) | -15.20 (1.11) | -16.96 (1.11)
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Longitudinal analysis to assess the average treatment effect over 48 months with visits at 6, 12, 18, 24, 30, 36, 42 and 48 months using all available data; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — p-value adjusted for 6 treatment group comparisons; Mixed effects model assuming data missing at random, adjusted for medical center as a random effect and for the baseline outcome score; Mean Difference (Net) = 3.15, 95% CI 2-sided [0.92 to 5.39] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.40, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.98, 95% CI 2-sided [-0.24 to 4.20] — Mean difference is the least squares mean changes from baseline for the memantine group minus the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.49, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.76, 95% CI 2-sided [-0.48 to 4.00] — Mean difference is the least squares mean changes from baseline for the vitamin E + memantine group minus the placebo group
Statistical Analysis 4: Comparison: Vitamin E vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.39, 95% CI 2-sided [-3.63 to 0.85] — Mean difference is the least squares mean changes from baseline for the vitamin E + memantine group minus the vitamin E group
Statistical Analysis 5: Comparison: Memantine vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.85, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.22, 95% CI 2-sided [-2.44 to 2.01] — Mean difference is the least squares mean changes from baseline for the vitamin E + memantine group minus the memantine group
Statistical Analysis 6: Comparison: Vitamin E vs Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.18, 95% CI 2-sided [-1.04 to 3.39] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the memantine group

2. Secondary Outcome: Dependence Scale: Time to Event Analysis (Increase of of One Dependence Level)
Description: The Dependence Scale assesses the level of assistance needed by patients with Alzheimer's disease for activities of daily living. The scale yields six levels of dependence: no assistance required (Level 0); requires occasional reminders (Level 1); requires frequent reminders and/or help with household chores (Level 2); needs daily supervision (Level 3); needs to be dressed, toileted or fed (Level 4); needs to be transferred, diapered or tube fed (Level 5).
Time Frame: Every 6 months to a maximum of 4 years
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Number; unit: participants
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 140 | 142 | 139 | 140
participants | 80 | 87 | 87 | 79
Statistical Analysis 1: Comparison: Vitamin E vs Memantine vs Vitamin E + Memantine vs Placebo; Test type: Superiority or Other; p = 0.69, Log Rank — p- value is unadjusted for multiple comparisons because its a 3 degrees of freedom test for any treatment group differences; 3 degrees of freedom test

3. Primary Outcome: Mini-Mental State Examination Change From Baseline
Description: The Mini-Mental State Examination (MMSE) briefly and objectively assess cognitive status in psychiatric patients with cognitive impairment. The MMSE questions are grouped into seven categories, each representing a different cognitive domain. The MMSE yields a total score that ranges from 0 for a patient who gives no correct response to a score of 30 for a patient who makes no errors. Outcome analysis is average least square means change from baseline.
Time Frame: 6, 12, 18, 24, 30, 36, 42 and 48 months minus baseline
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 136 | 140 | 136 | 137
units on a scale
  6 months minus baseline | -0.35 (0.29) | -0.24 (0.28) | -0.20 (0.29) | -0.34 (0.29)
  12 months minus baseline | -0.95 (0.34) | -1.09 (0.34) | -0.65 (0.34) | -1.39 (0.35)
  18 months minus baseline | -2.00 (0.44) | -2.62 (0.45) | -1.22 (0.44) | -2.21 (0.45)
  24 months minus baseline | -2.62 (0.52) | -3.44 (0.54) | -2.29 (0.53) | -2.90 (0.55)
  30 months minus baseline | -3.67 (0.61) | -3.79 (0.63) | -3.16 (0.61) | -3.26 (0.65)
  36 months minus baseline | -4.97 (0.74) | -4.26 (0.78) | -3.69 (0.73) | -3.87 (0.79)
  42 months minus baseline | -4.84 (0.79) | -4.59 (0.80) | -3.80 (0.74) | -4.68 (0.83)
  48 months minus baseline | -5.26 (0.94) | -5.98 (0.98) | -5.70 (0.91) | -5.42 (1.02)
  Average change from baseline | -2.97 (0.33) | -3.05 (0.33) | -2.80 (0.33) | -3.16 (0.33)
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.54 to 0.92] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.61 to 0.84] — Mean difference is the least squares mean changes from baseline for the memantine group minus the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.37, 95% CI 2-sided [-0.36 to 1.10] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Vitamin E vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.17, 95% CI [-0.56 to 0.90] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Memantine vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.47 to 0.98] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Vitamin E vs Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.65 to 0.80] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the memantine group

4. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) Change From Baseline
Description: The Alzheimer's Disease Assessment Scale (ADAS) is a 21-item scale designed to assess the severity of cognitive and non-cognitive behavioral impairments in patients with Alzheimer's disease. The cognitive portion of the scale (ADAS-cog) consists of 11 items to assess memory, language, and praxis functions. The ADAS-cog total score ranges from 0 (no errors) to 70 (severe cognitive impairment). Outcome analysis is average least square means change from baseline.
Time Frame: 6, 12, 18, 24, 30, 36, 42 and 48 months minus baseline
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 135 | 140 | 136 | 137
units on a scale
  6 months minus baseline | 1.38 (0.63) | 1.11 (0.62) | 1.53 (0.63) | 3.04 (0.63)
  12 months minus baseline | 2.40 (0.72) | 3.32 (0.72) | 2.48 (0.72) | 4.26 (0.74)
  18 months minus baseline | 4.34 (0.91) | 5.69 (0.91) | 3.46 (0.90) | 6.04 (0.92)
  24 months minus baseline | 4.32 (1.10) | 6.73 (1.12) | 5.76 (1.11) | 6.71 (1.15)
  30 months minus baseline | 7.87 (1.31) | 7.64 (1.34) | 5.85 (1.30) | 8.90 (1.38)
  36 months minus baseline | 9.00 (1.53) | 8.31 (1.60) | 8.26 (1.50) | 10.77 (1.63)
  42 months minus baseline | 10.35 (1.60) | 8.24 (1.64) | 7.97 (1.51) | 10.61 (1.69)
  48 months minus baseline | 10.73 (1.87) | 11.74 (1.97) | 9.70 (1.82) | 10.85 (2.04)
  Average change from baseline | 5.97 (0.70) | 6.38 (0.70) | 6.13 (0.71) | 7.78 (0.70)
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.80, 95% CI 2-sided [-3.28 to -0.33] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.25, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.39, 95% CI 2-sided [-2.85 to 0.07] — Mean difference is the least squares mean changes from baseline for the memantine group minus the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.65, 95% CI 2-sided [-3.12 to -0.17] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Vitamin E vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-1.32 to 1.63] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Memantine vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.26, 95% CI 2-sided [-1.72 to 1.21] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Vitamin E vs Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.41, 95% CI 2-sided [-1.88 to 1.06] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the memantine group

5. Primary Outcome: Neuropsychiatric Inventory Change From Baseline
Description: The Neuropsychiatric Inventory (NPI) assesses psychological and behavioral problems in patients with dementia. For each of twelve domains, there are four scores: frequency, severity, total frequency x severity, and caregiver distress. The frequency x severity total scores from each domain are summed for an overall total score that ranges from 0 to 144. The total caregiver distress scores are also summed for an overall total caregiver distress score that ranges from 0 to 60. The secondary endpoint for the trial will be the overall frequency times severity total score. Outcome analysis is average least square means change from baseline.
Time Frame: 6, 12, 18, 24, 30, 36, 42 and 48 months minus baseline
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 140 | 142 | 139 | 140
units on a scale
  6 months minus baseline | -1.24 (1.07) | -0.20 (1.06) | -0.47 (1.08) | 0.46 (1.07)
  12 months minus baseline | -1.04 (1.21) | 0.31 (1.22) | -0.17 (1.22) | 1.08 (1.24)
  18 months minus baseline | 0.93 (1.40) | 1.18 (1.43) | 0.41 (1.41) | 4.06 (1.44)
  24 months minus baseline | 2.16 (1.74) | 4.29 (1.79) | 1.98 (1.77) | 3.59 (1.84)
  30 months minus baseline | 3.21 (1.70) | 2.62 (1.71) | 2.16 (1.71) | 1.66 (1.81)
  36 months minus baseline | 2.15 (1.97) | 3.24 (2.07) | 2.79 (1.95) | 0.60 (2.16)
  42 months minus baseline | 0.81 (2.64) | 3.63 (2.75) | 1.85 (2.54) | 3.64 (2.89)
  48 months minus baseline | -0.60 (2.53) | 2.79 (2.60) | 5.14 (2.54) | 0.30 (2.79)
  Average change from baseline | 0.79 (1.00) | 1.87 (1.00) | 1.79 (1.00) | 2.26 (1.01)
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.46, 95% CI 2-sided [-3.55 to 0.63] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.39, 95% CI 2-sided [-2.47 to 1.70] — Mean difference is the least squares mean changes from baseline for the memantine group minus the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.47, 95% CI 2-sided [-2.57 to 1.63] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Vitamin E vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.99, 95% CI 2-sided [-1.09 to 3.07] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Memantine vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-2.16 to 1.99] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Vitamin E vs Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.08, 95% CI 2-sided [-3.14 to 0.99] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the memantine group

6. Primary Outcome: Caregiver Activity Survey Change From Baseline
Description: The Caregiver Activity Survey (CAS) was developed to measure the time caregivers spend aiding Alzheimer patients with their day-to-day activities. The CAS consists of six items that ask for an estimate in hours and minutes of the time that the caregiver spent during the previous 24 hours performing these particular activities. The six CAS items are as follows: 1) communication with the person, 2) using transportation, 3) dressing, 4) eating, 5) looking after one's appearance, and 6) supervising the person. The more caregiving hours the worse the patient's functioning level. Outcome analysis is average least square means change from baseline.
Time Frame: 6, 12, 18, 24, 30, 36, 42 and 48 months minus baseline
Population: Intention-to-treat analysis that includes all participants with baseline and at least one follow-up measurement.
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 140 | 142 | 139 | 140
hours per day
  6 months minus baseline | -0.93 (0.82) | 0.99 (0.81) | 1.08 (0.83) | 1.20 (0.82)
  12 months minus baseline | -0.18 (1.00) | 2.72 (1.01) | 1.39 (1.01) | 1.89 (1.04)
  18 months minus baseline | 2.12 (1.20) | 3.77 (1.22) | 2.69 (1.20) | 3.16 (1.23)
  24 months minus baseline | 1.60 (1.09) | 3.06 (1.13) | 2.82 (1.11) | 3.45 (1.16)
  30 months minus baseline | 4.14 (1.22) | 5.22 (1.25) | 3.41 (1.24) | 4.36 (1.32)
  36 months minus baseline | 7.69 (2.30) | 5.72 (2.43) | 4.90 (2.24) | 10.68 (2.51)
  42 months minus baseline | 4.95 (1.81) | 9.46 (1.89) | 5.48 (1.73) | 10.62 (1.99)
  48 months minus baseline | 10.17 (2.74) | 9.27 (2.80) | 13.80 (2.74) | 12.17 (3.03)
  Average change from baseline | 3.35 (0.78) | 5.52 (0.78) | 5.00 (0.78) | 5.14 (0.79)
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.79, 95% CI 2-sided [-3.35 to -0.23] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.38, 95% CI 2-sided [-1.18 to 1.94] — Mean difference is the least squares mean changes from baseline for the memantine group minus the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-1.70 to 1.42] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Vitamin E vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.65, 95% CI 2-sided [0.11 to 3.19] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Memantine vs Vitamin E + Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.52, 95% CI 2-sided [-2.07 to 1.02] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Vitamin E vs Memantine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — p-value is adjusted for 6 treatment group comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.17, 95% CI 2-sided [-3.71 to -0.63] — Mean difference is the least squares mean changes from baseline for the vitamin E group minus the memantine group

7. Other Pre Specified Outcome: All-cause Mortality
Description: Survival analysis of death from any cause.
Time Frame: up to 4 years
Population: Intention-to-treat analysis that includes all randomized participants.
Measure: Number; unit: participants
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Number analyzed (Participants) | 152 | 155 | 154 | 152
participants | 26 | 39 | 32 | 31
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.31, Log Rank — p-value is unadjusted for multiple comparisons; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.67 to 1.13] — Hazard ratio is for vitamin E group relative to the placebo group
Statistical Analysis 2: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.47, Log Rank — p-value is unadjusted for multiple comparisons; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.91 to 1.24] — Hazard ratio is for the memantine group relative to the placebo group
Statistical Analysis 3: Comparison: Vitamin E + Memantine vs Placebo; Test type: Superiority or Other; p = 0.80, Log Rank — p-value is unadjusted for multiple comparisons; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.57 to 1.54] — Hazard ratio is for the vitamin E + memantine group relative to the placebo group

ADVERSE EVENTS:
Arm/Group | Vitamin E | Memantine | Vitamin E + Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 82/152 | 84/155 | 83/154 | 95/152
Other Adverse Events (participants affected / at risk) | 91/152 | 97/155 | 90/154 | 89/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (N=152) | Memantine (N=155) | Vitamin E + Memantine (N=154) | Placebo (N=152)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (5)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (8) | 2 (2) | 4 (5) | 5 (7)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (7) | 5 (5) | 3 (3) | 4 (5)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1) | 3 (5) | 3 (4)
Complication of device insertion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 3 (5) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (11) | 8 (9) | 15 (15) | 5 (5)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sporotrichosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 8 (8) | 7 (13) | 4 (5)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (17) | 14 (16) | 12 (14) | 15 (18)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulation factor decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain mass (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cerebral amyloid angiopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Dementia Alzheimer's type (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (5)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Parasomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 3 (3) | 2 (2) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respite care (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Arterial bypass operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Drug detoxification (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospice care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 2 (4) | 1 (2) | 1 (1)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) — Sum of all adverse event terms in the Blood and Lymphatic Disorders System Organ Class
Cardiac Disorders (Cardiac disorders) | 19 (30) | 16 (23) | 19 (21) | 20 (26) — Sum of all adverse event terms in the Cardiac Disorders System Organ Class
Gastrointestinal Disorders (Gastrointestinal disorders) | 13 (13) | 14 (18) | 12 (13) | 8 (10) — Sum of all adverse event terms in the Gastrointestinal Disorders System Organ Class
General Disorders (General disorders) | 9 (9) | 7 (8) | 8 (10) | 14 (15) — Sum of all adverse event terms in the General Disorders System Organ Class
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) — Sum of all adverse event terms in the Hepatobiliary Disorders System Organ Class
Infections (Infections and infestations) | 19 (29) | 23 (31) | 31 (44) | 11 (13) — Sum of all adverse event terms in the Infections and Infestations System Organ Class
Injury or Procedural Complications (Injury, poisoning and procedural complications) | 18 (22) | 15 (18) | 15 (17) | 18 (21) — Sum of all adverse event terms in the Injury, Poisoning and Procedural Complications System Organ Class
Investigations (Investigations) | 2 (2) | 2 (2) | 4 (4) | 1 (1) — Sum of all adverse event terms in the Investigations System Organ Class
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 3 (4) | 7 (7) | 7 (9) | 6 (6) — Sum of all adverse event terms in the Matabolism and Nutrition Disorders System Organ Class
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (8) | 4 (6) | 6 (6) — Sum of all adverse event terms in the Neoplasm System Organ Class
Nervous System Disorders (Nervous system disorders) | 12 (15) | 15 (18) | 17 (18) | 19 (21) — Sum of all adverse event terms in the Nervous System Disorders System Organ Class
Psychiatric Disorders (Psychiatric disorders) | 8 (10) | 10 (10) | 5 (7) | 5 (5) — Sum of all adverse event terms in the Psychiatric Disorders System Organ Class
Renal and Urinary Disorders (Renal and urinary disorders) | 2 (2) | 5 (5) | 4 (4) | 6 (6) — Sum of all adverse event terms in the Renal and Urinary Disorders System Organ Class
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 9 (11) | 7 (8) | 11 (17) — Sum of all adverse event terms in the Respiratory Disorders System Organ Class
Skin Disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) — Sum of all adverse event terms in the Skin Disorders System Organ Class
Social Circumstances (Social circumstances) | 1 (2) | 1 (1) | 0 (0) | 3 (3) — Sum of all adverse event terms in the Social Circumstances System Organ Class
Surgical and Medical Procedures (Surgical and medical procedures) | 9 (10) | 5 (7) | 5 (6) | 5 (6) — Sum of all adverse event terms in the Surgical and Medical Procedures System Organ Class
Vascular Disorders (Vascular disorders) | 4 (4) | 5 (6) | 6 (9) | 6 (6) — Sum of all adverse event terms in the Vascular Disorders System Organ Class
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (N=152) | Memantine (N=155) | Vitamin E + Memantine (N=154) | Placebo (N=152)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Refraction disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 4 (8) | 8 (8) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (2) | 2 (2) | 3 (3) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (6) | 6 (7) | 2 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Drug dose omission (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Drug prescribing error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exposure to chemical pollution (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 31 (58) | 28 (39) | 37 (65) | 31 (48)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood albumin abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Blood homocysteine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Culture negative (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Full blood count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 4 (4) | 5 (5) | 3 (4) | 3 (3)
Prostatic specific antigen increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3) | 0 (0) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 7 (8) | 5 (5) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Abnormal sleep-related event (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (2)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Social avoidant behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dialysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Emergency care (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No